CLINICAL TRIAL: NCT01703221
Title: A Phase III, Multicenter, Randomized, Placebo- and Sitagliptin-controlled, Parallel-group, Double-blinded Study and Subsequent Open-label, Extension Study to Assess the Safety and Efficacy of MK-3102 in Japanese Patients With Type 2 Diabetes Mellitis Who Have Inadequate Glycemic Control on Diet/Exercise Therapy
Brief Title: Omarigliptin (MK-3102) Clinical Trial - Placebo- and Sitagliptin-Controlled Monotherapy Study in Japanese Patients With Type 2 Diabetes Mellitus (MK-3102-020)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3102-020; 132239 (Registry Identifier: JAPIC-CTI)
Record Dates: First submitted 2012-10-05; First posted 2012-10-10 (Estimated); Results first posted 2015-10-29 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — 2-(2,5-difluorophenyl)-5-(2-(methylsulfonyl)-2,6-dihydropyrrolo(3,4-c)pyrazol-5(4H)-yl)tetrahydro-2H-pyran-3-amine; Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Omarigliptin 25 mg (Phase A+B) (Experimental): Omarigliptin 25 mg once weekly for 52 weeks (Phase A + B)
  Interventions: Drug: Omarigliptin; Drug: Placebo to sitagliptin
- Sitagliptin (Phase A) switching to Omarigliptin (Phase B) (Active Comparator): Sitagliptin 50 mg once daily for 24 weeks (Phase A) switching to omarigliptin 25 mg once weekly for 28 weeks (Phase B)
  Interventions: Drug: Omarigliptin; Drug: Sitagliptin; Drug: Placebo to omarigliptin
- Placebo (Phase A) switching to Omarigliptin (Phase B) (Placebo Comparator): Placebo for 24 weeks (Phase A) switching to omarigliptin 25 mg once weekly for 28 weeks (Phase B)
  Interventions: Drug: Omarigliptin; Drug: Placebo to omarigliptin; Drug: Placebo to sitagliptin

INTERVENTIONS:
Drug: Omarigliptin — Omarigliptin (MK-3102) 25 mg capsule administered orally once weekly
Drug: Sitagliptin — Sitagliptin 50 mg tablet administered orally once daily
  Other Names: Januvia®
  Arms: Sitagliptin (Phase A) switching to Omarigliptin (Phase B)
Drug: Placebo to omarigliptin — Placebo to omarigliptin 25 mg capsule administered orally once weekly
  Arms: Placebo (Phase A) switching to Omarigliptin (Phase B); Sitagliptin (Phase A) switching to Omarigliptin (Phase B)
Drug: Placebo to sitagliptin — Placebo to sitagliptin 50 mg tablet administered orally once daily
  Arms: Omarigliptin 25 mg (Phase A+B); Placebo (Phase A) switching to Omarigliptin (Phase B)

SUMMARY:
The purpose of this study is to assess the efficacy of omarigliptin 25 mg weekly (as monotherapy) compared with sitagliptin 50 mg daily and placebo, and the long term safety (up to 52 weeks) of omarigliptin 25 mg weekly. The primary hypotheses are that after 24 weeks: 1) Omarigliptin 25 mg weekly provides a greater reduction from baseline in glycosylated hemoglobin (HbA1c) compared with placebo, and 2) The mean change from baseline in HbA1c in participants treated with omarigliptin 25 mg weekly is non-inferior compared with that in participants treated with sitagliptin 50 mg daily.

DETAILED DESCRIPTION:
The treatment period is composed of a 24-week double-blind period (Phase A) and a 28-week open-label period (Phase B). Participants will receive in Phase A: omarigliptin 25 mg once weekly, sitagliptin 50 mg once daily or placebo and in Phase B: omarigliptin 25 mg once weekly.

ELIGIBILITY:
Inclusion Criteria:

* Has type 2 diabetes mellitus

Exclusion Criteria:

* History of type 1 diabetes mellitus or a history of ketoacidosis
* History of any of the following medications: thiazolidinediones and/or insulin within 12 weeks prior to study participation, omarigliptin and/or sitagliptin anytime

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 414 (Actual)
Dates: Start 2012-10-24 (Actual); Primary Completion 2014-04-25 (Actual); Study Completion 2014-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Gantz I, Okamoto T, Ito Y, Okuyama K, O'Neill EA, Kaufman KD, Engel SS, Lai E; the Omarigliptin Study 020 Group. A randomized, placebo- and sitagliptin-controlled trial of the safety and efficacy of omarigliptin, a once-weekly dipeptidyl peptidase-4 inhibitor, in Japanese patients with type 2 diabetes. Diabetes Obes Metab. 2017 Nov;19(11):1602-1609. doi: 10.1111/dom.12988. Epub 2017 Jul 6. PMID 28449368
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=3102-020&kw=3102-020&tab=access

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Forty-eight sites in Japan received IRB approval and were shipped clinical supplies in this study and randomized at least one participant. One hundred and seventeen participants were not randomized; the most common reason for participants not being randomized was screen failure.
Pre-assignment Details: In Phase A, participants were randomized to receive either omarigliptin 25 mg once weekly, sitagliptin 50 mg once daily or placebo for 24 weeks in a blinded manner. In Phase B, all participants received open-label omarigliptin 25 mg once weekly for 28 weeks.
Groups:
- Omarigliptin (Phase A+B): Omarigliptin 25 mg once weekly for 52 weeks (Phase A + B)
Period: Phase A (Up to 24 Weeks)
Arm/Group | Omarigliptin (Phase A+B) | Sitagliptin (Phase A) Switching to Omarigliptin (Phase B) | Placebo (Phase A) Switching to Omarigliptin (Phase B)
Started | 166 | 165 | 83
Completed | 159 | 161 | 80
Not Completed | 7 | 4 | 3
Not completed — Adverse Event | 2 | 4 | 0
Not completed — Lack of Efficacy | 2 | 0 | 1
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 1
Period: Phase B - (Week 25 to 52)
Arm/Group | Omarigliptin (Phase A+B) | Sitagliptin (Phase A) Switching to Omarigliptin (Phase B) | Placebo (Phase A) Switching to Omarigliptin (Phase B)
Started | 159 | 161 | 80
Completed | 143 | 147 | 75
Not Completed | 16 | 14 | 5
Not completed — Withdrawal by Subject | 2 | 1 | 0
Not completed — Adverse Event | 2 | 3 | 2
Not completed — Lack of Efficacy | 12 | 10 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Omarigliptin (Phase A+B) | Sitagliptin (Phase A) Switching to Omarigliptin (Phase B) | Placebo (Phase A) Switching to Omarigliptin (Phase B) | Total
Number analyzed (Participants) | 166 | 165 | 83 | 414
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60 (11) | 60 (9) | 61 (9) | 60 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 50 | 26 | 138
  Male | 104 | 115 | 57 | 276

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline for Hemoglobin A1c (HbA1c) at Week 24
Description: HbA1C is blood marker used to report average blood glucose levels over prolonged periods of time and is reported as a percentage (%). Change in A1C following 24 weeks of therapy (i.e., A1C at Week 24 minus A1C at baseline).
Time Frame: Baseline and Week 24
Population: The Full Analysis Set (FAS) consisted of all randomized participants who had at least one study drug and had a baseline or post-randomization measurement for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent HbA1c
Groups:
- Omarigliptin (Phase A): Omarigliptin 25 mg once weekly for 24 weeks (Phase A)
- Sitagliptin (Phase A): Sitagliptin 50 mg once daily for 24 weeks (Phase A)
- Placebo (Phase A): Placebo for 24 weeks (Phase A)
Arm/Group | Omarigliptin (Phase A) | Sitagliptin (Phase A) | Placebo (Phase A)
Number analyzed (Participants) | 166 | 164 | 82
Percent HbA1c | -0.66 [-0.76 to -0.57] | -0.65 [-0.74 to -0.55] | 0.13 [-0.00 to 0.27]
Statistical Analysis 1: Comparison: Omarigliptin (Phase A) vs Placebo (Phase A); Test type: Superiority or Other; p < 0.001, Constrained longitudinal analysis; Terms for treatment, prior oral antihyperglycemic agent (AHA), time, time by: treatment, prior AHA therapy status, and treatment by prior AHA status; Difference in the least squares means = -0.80, 95% CI 2-sided [-0.96 to -0.63]
Statistical Analysis 2: Comparison: Sitagliptin (Phase A) vs Placebo (Phase A); Test type: Superiority or Other; p < 0.001, Constrained longitudinal analysis; Terms for treatment, prior AHA therapy status (yes/no), time, and time by: treatment, prior AHA therapy status, and treatment by prior AHA status; Difference in the least squares means = -0.78, 95% CI 2-sided [-0.94 to -0.61]
Statistical Analysis 3: Comparison: Omarigliptin (Phase A) vs Sitagliptin (Phase A); Test type: Non-Inferiority or Equivalence — Omarigliptin will be considered non-inferior to sitagliptin if the upper bound of the two-sided 95% confidence interval of the between-treatment difference in least squares means for change from baseline in HbA1c at Week 24 (omarigliptin minus sitagliptin) is not more than 0.3% (non-inferiority margin); p = 0.792, Constrained longitudinal analysis; [statistical method as in outcome 1, analysis 2]; Difference in the least squares means = -0.02, 95% CI 2-sided [-0.15 to 0.12]

2. Primary Outcome: Percentage of Participants Who Experienced at Least One Adverse Event During Phase A
Description: An adverse event (AE) is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study.
Time Frame: Up to 24 weeks
Population: All Subjects as Treated (ASaT) population consisted of all randomized participants who received at least one study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Omarigliptin (Phase A) | Sitagliptin (Phase A) | Placebo (Phase A)
Number analyzed (Participants) | 166 | 164 | 82
Percentage of participants | 50.0 | 49.4 | 65.9

3. Primary Outcome: Percentage of Participants Who Experienced at Least One Adverse Event During the Overall Study
Description: An AE is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study. These results represent the accrual of events over different treatment intervals: 52 weeks, omarigliptin (Phase A+B) defined as the double-blind period and open label extension period versus 28 weeks for the Sitagliptin (Phase A)→Omarigliptin (Phase B) and placebo (Phase A)→Omarigliptin (Phase B) group defined as the open-label extension period only.
Time Frame: Up to 52 weeks
Population: The ASaT Population included all randomized participants who received at least one study drug. Data was unavailable for 7 participants who discontinued the study in sitagliptin and placebo arms in Phase A.
Measure: Number; unit: Percentage of Participants
Groups:
- Omarigliptin (Phase B)-S: Omarigliptin 25 mg once weekly for 28 weeks (Phase B) after switching from sitagliptin
- Omarigliptin (Phase B)-P: Omarigliptin 25 mg once weekly for 28 weeks (Phase B) after switching from placebo
Arm/Group | Omarigliptin (Phase A+B) | Omarigliptin (Phase B)-S | Omarigliptin (Phase B)-P
Number analyzed (Participants) | 166 | 161 | 80
Percentage of Participants | 69.9 | 47.2 | 56.3

4. Primary Outcome: Percentage of Participants Who Discontinued From the Study Due to an Adverse Event During Phase A
Description: An AE is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study.
Time Frame: Up to 24 weeks
Population: The ASaT Population consisted of all randomized participants who received at least one study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Omarigliptin (Phase A) | Sitagliptin (Phase A) | Placebo (Phase A)
Number analyzed (Participants) | 166 | 164 | 82
Percentage of participants | 0.6 | 1.2 | 0

5. Primary Outcome: Percentage of Participants Who Discontinued From the Study Due to an Adverse Event During the Overall Study
Description: as for outcome 3
Time Frame: Up to 52 weeks
Population: The ASaT Population consisted of all randomized participants who received at least one study drug. Data was unavailable for 7 participants who discontinued the study in sitagliptin and placebo arms in Phase A.
Measure: Number; unit: Percentage of participants
Arm/Group | Omarigliptin (Phase A+B) | Omarigliptin (Phase B)-S | Omarigliptin (Phase B)-P
Number analyzed (Participants) | 166 | 161 | 80
Percentage of participants | 2.4 | 1.2 | 1.3

6. Secondary Outcome: Change From Baseline for 2-hour Post Meal Glucose (PMG) at Week 24
Description: Change from baseline at Week 24 is defined as PMG at Week 24 minus PMG at Week 0.
Time Frame: Baseline and Week 24
Population: The FAS Population consisted of all randomized participants who had at least one study drug and had a baseline or post-randomization measurement for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Omarigliptin (Phase A) | Sitagliptin (Phase A) | Placebo (Phase A)
Number analyzed (Participants) | 166 | 164 | 82
mg/dL | -42.38 [-49.53 to -35.23] | -45.24 [-52.31 to -38.16] | -5.48 [-15.13 to 4.17]
Statistical Analysis 1: Comparison: Omarigliptin (Phase A) vs Placebo (Phase A); Test type: Superiority or Other; p < 0.001, Constrained longitudinal analysis; [statistical method as in outcome 1, analysis 2]; Difference in the least squares means = -36.89, 95% CI 2-sided [-48.46 to -25.33]
Statistical Analysis 2: Comparison: Sitagliptin (Phase A) vs Placebo (Phase A); Test type: Superiority or Other; p < 0.001, Constrained longitudinal analysis; [statistical method as in outcome 1, analysis 2]; Difference in the least squares means = -39.76, 95% CI 2-sided [-51.28 to -28.23]
Statistical Analysis 3: Comparison: Omarigliptin (Phase A) vs Sitagliptin (Phase A); Test type: Superiority or Other; p = 0.555, Constrained longitudinal analysis; [statistical method as in outcome 1, analysis 2]; Difference in the least squares means = 2.86, 95% CI 2-sided [-6.67 to 12.39]

7. Secondary Outcome: Change From Baseline for Fasting Plasma Glucose (FPG) at Week 24
Description: Blood glucose was measured on a fasting basis. FPG is expressed as mg/dL. Blood was drawn at predose on Day 1 and after 24 weeks of treatment to determine change in plasma glucose levels (i.e., FPG at Week 24 minus FPG at baseline).
Time Frame: Baseline and Week 24
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Omarigliptin (Phase A) | Sitagliptin (Phase A) | Placebo (Phase A)
Number analyzed (Participants) | 166 | 164 | 82
mg/dL | -18.52 [-21.81 to -15.22] | -20.75 [-24.10 to -17.39] | -6.23 [-10.84 to -1.63]
Statistical Analysis 1: Comparison: Omarigliptin (Phase A) vs Placebo (Phase A); Test type: Superiority or Other; p < 0.001, Constrained longitudinal analysis; [statistical method as in outcome 1, analysis 2]; Difference in the least squares means = -12.28, 95% CI 2-sided [-17.78 to -6.78]
Statistical Analysis 2: Comparison: Sitagliptin (Phase A) vs Placebo (Phase A); Test type: Superiority or Other; p < 0.001, Constrained longitudinal analysis; [statistical method as in outcome 1, analysis 2]; Difference in the least squares means = -14.51, 95% CI 2-sided [-20.04 to -8.98]
Statistical Analysis 3: Comparison: Omarigliptin (Phase A) vs Sitagliptin (Phase A); Test type: Superiority or Other; p = 0.330, Constrained longitudinal analysis; [statistical method as in outcome 1, analysis 2]; Difference in the least squares means = 2.23, 95% CI 2-sided [-2.27 to 6.73]

ADVERSE EVENTS:
Time Frame: Phase A (up to 24 weeks), Phase B (Up to 28 weeks [Week 25 to 52]), Phase A+B (up to 52 weeks)
Description: The ASaT population was all randomized participants who received at least 1 study drug. Note: these AE results represent the accrual of AEs over different treatment intervals: 52 weeks, omarigliptin (Phase A+B): double-blind period (DBP) + open label extension period (OLEP) versus 24 weeks (DBP) or 28 weeks (OLEP) for all other study arms.
Groups:
- Omarigliptin (Phase A + B): Omarigliptin 25 mg once weekly for 52 weeks (Phase A + B)
Arm/Group | Omarigliptin (Phase A) | Sitagliptin (Phase A) | Placebo (Phase A) | Omarigliptin (Phase A + B) | Omarigliptin (Phase B)-S | Omarigliptin (Phase B)-P
Serious Adverse Events (participants affected / at risk) | 3/166 | 3/164 | 0/82 | 6/166 | 2/161 | 0/80
Other Adverse Events (participants affected / at risk) | 21/166 | 18/164 | 25/82 | 45/166 | 22/161 | 17/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omarigliptin (Phase A) (N=166) | Sitagliptin (Phase A) (N=164) | Placebo (Phase A) (N=82) | Omarigliptin (Phase A + B) (N=166) | Omarigliptin (Phase B)-S (N=161) | Omarigliptin (Phase B)-P (N=80)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Limb traumatic amputation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sick sinus syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omarigliptin (Phase A) (N=166) | Sitagliptin (Phase A) (N=164) | Placebo (Phase A) (N=82) | Omarigliptin (Phase A + B) (N=166) | Omarigliptin (Phase B)-S (N=161) | Omarigliptin (Phase B)-P (N=80)
Nasopharyngitis (Infections and infestations) | 21 (24) | 18 (22) | 25 (27) | 45 (58) | 22 (30) | 17 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results.